CLINICAL TRIAL: NCT02583945
Title: Effect of a Kidney Bundle on the Occurence of Postoperative Acute Kidney Injury in Patients at Risk
Brief Title: Prevention of Postoperative Acute Kidney Injury
Acronym: PrevenAKI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study medication without approval and stop of financial support
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. Christian Wunder, Vice chair and leading senior physician, Wuerzburg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 022015
Record Dates: First submitted 2015-09-23; First posted 2015-10-22 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; hemodynamic stabilisation; nephrotoxic medication
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kidney treatment bundle (KDIGO) (Experimental): Consequent postoperative application of a kidney treatment bundle: Protocol based hemodynamic optimization and monitoring, regular screening of creatinine in serum and of urine output, no use of potential nephrotoxic medication and normoglycemia.
  Interventions: Procedure: kidney treatment bundle (KDIGO)

INTERVENTIONS:
Procedure: kidney treatment bundle (KDIGO) — Application of the measures of the kidney treatment bundle.

SUMMARY:
Postoperative acute kidney injury (AKI) refers to increased mortality and morbidity in patients after non-cardiac surgery. The Kidney Disease Improving Global Outcomes (KDIGO)-guidelines recommend a bundle of procedures to prevent the occurrence of AKI: A protocol for the improvement of the hemodynamic situation and a standardized proceeding in hemodynamic monitoring, consequent avoidance of nephrotoxic substances, regular measurement of creatinine and urine output, as well as normoglycemia. The primary goal is to determine if the consequent application of the KDIGO-bundle leads to a prevention of the occurrence of AKI in patients at risk after non-cardiac surgery.

DETAILED DESCRIPTION:
All patients included in the study will be treated with the KDIGO-bundle (hemodynamic stabilization, avoidance of nephrotoxic substances, normoglycemia and measurement of creatinine in serum and urine output). 12 h, 24h as well as on day 2, 3, 5 and 10 after admission on ICU the occurence of AKI (according to KDIGO) will be assessed.

ELIGIBILITY:
Inclusion criteria:

* Age > 65 years
* chronic kidney disease
* diabetes mellitus, chronic heart, lung or liver disease
* hemodynamic instability (intra and/or post-operative)
* trauma, burn injury, major surgery, usage of x-ray contrast and sepsis.

Exclusion criteria:

* Age < 18 years
* pregnancy
* kidney graft recipient
* chronic renal disease with or without renal replacement therapy and cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative AKI | until day 5 after surgery
  AKI according to KDIGO definition

SECONDARY OUTCOMES:
Intensive care unit mortality | 28 days and 90 days after surgery
hospital mortality | up to 100 days after surgery
usage of renal replacement therapy (hours) | up to 30 days after surgery
length of invasive respirator therapy (hours) | up to 30 days after surgery
creatinine in serum | 12 hours, day 2, 3, 5 and 10 after surgery
urine output (total ml) | after 12 hours, on day 2 (in 24hour), 3 (in 24hour), 5 (in 24hour) and 10 (in 24hour) after surgery
length of hospital stay | up to 100 days after surgery
length of ICU stay | up to 100 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wunder, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- University Hospital Wuerzburg, Dep. of Anesthesiology, Würzburg, Germany